CLINICAL TRIAL: NCT06321029
Title: Electronic Diabetes Tune-Up Group (eDTU) for African Americans: A Pragmatic Trial Phase 2
Brief Title: Electronic Diabetes Tune-Up Group (eDTU) for African Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Mary de Groot, Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-22-ICTSHD-44
Record Dates: First submitted 2024-01-04; First posted 2024-03-20 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Complications
Keywords: Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Single group waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm waitlist control (Experimental): The initial assessment will take place at the time of study enrollment (T1). Participants will be offered a choice of assignment to either the eDTU (online Diabetes Tune-Up Group intervention participation) or iDTU (in-person Diabetes Tune-Up Group intervention participation) series. After a 3-month waiting period, participants will complete baseline assessment (T2). The group intervention will then take place over the next 6 to 8 weeks. Immediately following completion of the intervention, participants will complete surveys (T3). A final assessment will be completed 3 months after baseline, approximately 4 to 6 weeks following the completion of the intervention (T4).
  The participant will participate in one series of the DTU intervention either, in person or online, at the participant's choosing. The intervention will take place over the course of 6 to 8 weeks. Participants will wear their continuous glucose monitor throughout the course of the intervention.
  Interventions: Behavioral: Diabetes Tune-Up Group

INTERVENTIONS:
Behavioral: Diabetes Tune-Up Group — The eDTU and iDTU interventions will consist of 6 weekly group sessions lasting 90 minutes per session offered over a 6-8 week period. Each series will be co-facilitated by one diabetes care and education specialist and one behavioral health interventionist. Enrollment in each series will consist of 4-10 patients per group. The intervention components integrate key strategies that have been demonstrated to be effective in previous studies: motivational interviewing and introduction to stages of change; diabetes education; cognitive behavioral therapy with a particular emphasis on identification of cognitive distortions, thought stopping and cognitive reframing; emotional regulation; social support and miscarried helping; and behavioral strategies to support diabetes self-management. Each session will involve a psychoeducational portion, group discussion, and take-home assignments to be completed between sessions.

SUMMARY:
The primary aims of this study are:

1. To test the acceptability and feasibility of the electronic DTU intervention (eDTU) that has been adapted for cultural relevance and online delivery compared to waitlist control and the in-person DTU (iDTU). The hypothesis is that the adapted intervention will be culturally acceptable (by participant satisfaction scores) and well-subscribed (intervention attendance rates).
2. To test differences in diabetes distress and A1c change scores between intervention (changes in T2 to T4) and waitlist control (change in T1 to T2) by intervention group (eDTU vs. waitlist control; iDTU vs. waitlist control). The hypothesis is that both the eDTU and iDTU groups will show significant improvements in diabetes distress and A1c compared to waitlist control. In order to conserve sample size and budget, participants in each intervention group will serve as their own waitlist control.

Secondary Objective. The secondary aim of the study is to evaluate changes in depressive symptoms, diabetes self-efficacy, and general and diabetes-specific quality of life in intervention (T2-T3 & T4) compared to waitlist control (T1-T2). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (T2-T3 & T4). The hypothesis is that both groups will show comparable improvements in diabetes distress and A1c.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Self-identified Black or African American female
* Type 2 diabetes diagnosis ≥ 1 year
* A1c ≥ 7.0% in the past year per medical record or patient report
* DDS-17 score ≥ 2.0 at screening
* Active email address

Exclusion Criteria:

* Limited English language proficiency
* Presence of serious mental health disorder (e.g., psychotic disorders or severe mood disorders with suicidal ideation)
* Diagnosis of a major acute medical condition (e.g., myocardial infarction, stroke, cardiac rehabilitation, stage 3 or stage 4 cancer diagnoses) within the last three months
* Initiation of new medical treatment regimens (e.g., chemotherapy) for acute medical diagnoses that would require the patient's primary attention

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress Scale-17 (DDS-17) | To test differences in DDS-17 change scores between intervention (changes in baseline to 3-month follow-up) and waitlist control (change in enrollment to baseline) by intervention group (eDTU vs. waitlist control; iDTU vs. waitlist control).
  Change in DDS-17 scores over time; scores range from 1 - 6 with higher scores indicating worse diabetes distress
HbA1c (A1c) | To test differences in A1c change scores between intervention (changes in baseline to 3-month follow-up) and waitlist control (change in enrollment to baseline) by intervention group (eDTU vs. waitlist control; iDTU vs. waitlist control).
  Change in A1c values over time
Acceptability of intervention (content and delivery modality) | Immediately following intervention
  Acceptability of electronic DTU intervention (eDTU) adapted for cultural relevance and online delivery compared to waitlist control and the in-person DTU (iDTU) using study-developed satisfaction questionnaire; scores can range from 15 - 75 with higher scores indicating greater participant satisfaction
Feasibility of intervention and delivery modality | During intervention (6-8 weeks)
  Feasibility of electronic DTU intervention (eDTU) adapted for online delivery compared to the in-person DTU (iDTU) using participant attendance to intervention sessions; attendance will range from 1 to 6 sessions

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Evaluate changes in depressive symptoms in intervention (baseline to 3-month follow-up) compared to waitlist control (enrollment to baseline). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (baseline -3mo f/u).
  Evaluate changes in depressive symptoms in intervention (baseline to 3-month follow-up) compared to waitlist control (enrollment to baseline). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (baseline & three-month follow-up); scores range from 0 - 27 with higher scores indicating more severe depression symptoms
Confidence in Diabetes Self-Care (CDSC) | Evaluate changes in diabetes self-efficacy in intervention (baseline to 3-month follow-up) compared to waitlist control (enrollment to baseline).
  Evaluate changes in diabetes self-efficacy in intervention (baseline to 3mo f/u) compared to waitlist control (T1-T2). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (T2-T3 & T4); scores ranges from 20 - 100 with higher scores indicative of greater patient belief in caring for their diabetes
Short Form-12 (SF-12) | Evaluate changes in general quality of life in intervention (baseline to 3mo f/u) compared to waitlist control (enrollment-baseline). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (baseline to 3mo f/u).
  Evaluate changes in general quality of life in intervention (baseline to 3mo f/u) compared to waitlist control (T1-T2). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (T2-T3 & T4); Items are divided into 2 subscales, the Physical Component and Mental Component scores, total item and subscale scores are converted to a 100-point scale, with higher scores indicating better functioning.
Diabetes Therapy-Related Quality of Life Questionnaire | Evaluate changes in diabetes-specific quality of life in intervention (baseline to 3mo f/u) compared to waitlist control (enrollment-baseline). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (baseline to 3mo f/u).
  Evaluate changes in diabetes-specific quality of life in intervention (baseline to 3mo f/u) compared to waitlist control (T1-T2). An exploratory aim will be to compare changes in eDTU to the iDTU pre/post intervention (T2-T3 & T4); scores range from 17 - 68 with higher scores reflecting greater diabetes-specific quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will submit a Material Transfer Agreement form to the National Institute for Diabetes and Digestive and Kidney Diseases (NIDDK) Repository to seek approval for depositing de-identified data collected from all time points of the study.
Supporting Information: Study Protocol, ICF
Time Frame: Within 18 months of completion of the project

REFERENCES:
- [Background] de Groot M, Myers BA, Baker L, Daily E, Cavaghan M. The Diabetes Tune-Up Group: A Multidisciplinary Approach to Improve Diabetes Distress and A1C Among Adults With Type 1 and Type 2 Diabetes. Sci Diabetes Self Manag Care. 2023 Apr;49(2):150-162. doi: 10.1177/26350106231151405. Epub 2023 Jan 20. PMID 36661126